CLINICAL TRIAL: NCT00291538
Title: Comparison of Pharmacokinetics and Pharmacodynamics of Subcutaneous Versus Intravenous Administration of Bortezomib in Patients With Multiple Myeloma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BRD/05/9-B
Record Dates: First submitted 2006-02-10; First posted 2006-02-14 (Estimated); Last update posted 2009-02-04 (Estimated); Status verified 2009-02

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Bortezomib

INTERVENTIONS:
Drug: bortezomib

SUMMARY:
In this open-label randomised phase I trial, bortezomib will be administrated to 2 groups of 10 patients with MM who have inclusion criteria use the extended 2nd line indication, either intravenously (group 1 = 10 patients) or subcutaneously (group 2 = 10 patients). The schedule of administration of bortezomib will be the following : 1.3 mg per square meter of body-surface area twice weekly for 2 weeks, followed by 1 week without treatment, for up to eight cycles, either IV (group 1) or SC (group 2).

The primary objective is to characterize the pharmacokinetics of the 2 routes of administration.

The secondary objectives are to characterize the pharmacodynamics (20S proteasome inhibition in whole blood), toxicity, including cardiac safety, and efficacy of the 2 routes of administration.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of MM according to the SWOG criteria (annex I)
* symptomatic MM stage II or III according to Durie-Salmon staging system (annex II) or stage I with one symptomatic osteolytic lesion
* with progressive disease after at least one prior therapy and who have already undergone or are unsuitable for bone marrow transplantation
* with measurable levels of paraprotein in the serum (> 1g/dl) or in the urine (> 0.2g/24h)
* age < 75 years
* able to understand and to given an informed consent
* male, female without childbearing potential or negative urine pregnancy test within 72 hours prior to beginning the treatment. Women of childbearing potential must be following adequate contraceptive measures. Men must agree to use an acceptable method of contraception (for themselves or female partners) for the duration of the study
* no active systemic infection. In the presence of any active systemic infection, adequate broad-spectrum or organism-specific antibiotic coverage must be administered. Patients must be afebrile with stable vital signs while receiving antibiotics for at least 48 hours prior to beginning the treatment with Bortezomib.
* Each subject will weigh ³50 kg and have a body mass index (BMI) of £30 kg/m2 (see annex V for BMI formula).

Exclusion Criteria:

* life expectancy < 2 months
* ECOG performance status > 2 (annex III)
* proven amyloidosis
* positive HIV serology
* antecedents of severe psychiatric disease
* > NCI grade 2 peripheral neuropathy (Annex IV)
* History of clinically relevant cardiac disease, including prior myocardial infarction, prior or existing heart failure, existing uncontrolled angina or clinically significant pericardial disease Evidence of arrhythmia, 2nd degree or greater AV block or prolonged QTc interval (>0.45 seconds in males, >0.47 seconds in females) on screening ECG
* serum biochemical values as follow
* creatinine level > 200mmol/l
* bilirubin, transaminases or gGT > 3 the upper normal limit
* potassium, calcium or magnesium outside of upper or lower normal limits
* haematology values as follow
* platelet < 70x 109 /L within 14 days of enrollment
* absolute neutrophil count <1.0 x 109/L within 14 days of enrolment
* concomitant use of drugs able to modify QTc interval within 1 week prior to the first dose of bortezomib and during Cycle 1 (Annex VI)
* concomitant use of potent inhibitors or inducers of the cytochrome P450 (CYP) enzymes 3A and 2C19 within 1 week prior to the first dose of bortezomib and during Cycle 1 (see annex VII list of representative drugs).
* use of any experimental drugs within 30 days of baseline
* hypersensitivity to bortezomib, boron, or mannitol

Max Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2006-02; Primary Completion 2007-06 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
characterize the pharmacokinetics of the 2 routes of administration.

SECONDARY OUTCOMES:
characterize the pharmacodynamics (20S proteasome inhibition in whole blood),
toxicity, including cardiac safety,
efficacy of the 2 routes of administration.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Luc HAROUSSEAU, MD, Principal Investigator — Nantes UH
Locations (3):
- France (3):
  - Lille UH, Lille
  - Nancy UH, Nancy
  - Nantes UH, Nantes

REFERENCES:
- [Derived] Moreau P, Coiteux V, Hulin C, Leleu X, van de Velde H, Acharya M, Harousseau JL. Prospective comparison of subcutaneous versus intravenous administration of bortezomib in patients with multiple myeloma. Haematologica. 2008 Dec;93(12):1908-11. doi: 10.3324/haematol.13285. Epub 2008 Sep 2. PMID 18768528